CLINICAL TRIAL: NCT01676753
Title: A Phase 1b Trial of the Cyclin-dependent Kinase Inhibitor Dinaciclib in Combination With Pembrolizumab in Patients With Advanced Breast Cancer and Assessment of MYC Oncogene Overexpression
Brief Title: Phase 1b Trial of Dinaciclib With Pembrolizumab for Advanced Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jo Chien (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Jo Chien, UCSF Assistant Clinical Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16758; NCI-2018-01053 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2012-08-24; First posted 2012-08-31 (Estimated); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Advanced or Metastatic Breast Cancer; Triple Negative Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — dinaciclib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Dinaciclib, Pembrolizumab) (Experimental): Pembrolizumab will be administered on Day 1, every 3 weeks at a fixed dose of 200 mg IV. Dinaciclib will be administered D1 and D8 of a 21 day cycle by 2-hour intravenous infusion starting at Dose Level (DL) 1 of 12 mg/m^2. Further dose escalation cohorts are defined as follows: DL 2: 18 mg/m^2, DL 3: 25 mg/m^2, DL 4: 33 mg/m^2, and DL 5: 50 mg/m^2
  Interventions: Drug: Dinaciclib; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Dinaciclib — Given IV
  Other Names: SCH727965
Drug: Pembrolizumab — Given IV
  Other Names: Keytruda

SUMMARY:
The purpose of this trial is to determine the safety and tolerability (maximum tolerated dose (MTD)) of weekly dinaciclib in combination with pembrolizumab in patients with advanced breast cancer. Once this is defined, dose expansion will be performed at this MTD in patients with metastatic or locally advanced and unresectable triple negative breast cancer, to evaluate the efficacy of combined dinaciclib and pembrolizumab.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Define the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of dinaciclib

SECONDARY OBJECTIVE:

I. Evaluation of the preliminary efficacy of this combination using RECIST 1.1 and irRECIST.

EXPLORATORY OBJECTIVE:

I. Characterizing and correlating PDL-1 and MYC overexpression with clinical response.

OUTLINE:

This is an open-label phase Ib trial of weekly dinaciclib in combination pembrolizumab in participants with advanced triple negative breast cancer. Participants will undergo a single needle biopsy of a site of active disease prior to initiating treatment of Pembrolizumab and dinaciclib in 21 day cycles. The dose of dinaciclib will be escalated following a toxicity probability interval (TPI) design where dose-limiting toxicities (DLT) observed during the first cycle will be used to determine whether additional participants should be enrolled at the same, higher, or lower dose level. Treatment will continue until disease progression, intolerable toxicity, or participant withdraws consent. In the event of a complete response (CR), participants may elect to hold dinaciclib treatment and continue with pembrolizumab alone. At the time of radiographic disease progression, dinaciclib can be resumed at the same dose as at the time of discontinuation. Participants will be followed for 30 days after the last dose of treatment.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Histologically or cytologically documented, incurable, unresectable locally advanced, or metastatic breast cancer
2. Histologically documented metastatic or locally advanced unresectable breast cancer that is ER and progesterone receptor (PR) <10% expression and does not over-express Hormone Estrogen Receptor-Positive (HER2) protein (Immunohistochemistry (IHC) 0, 1+, or 2+ and Fluorescent in situ hybridization (FISH) <2.0)
3. Patient must consent to a biopsy of a site of disease unless the only site of disease is lung/pleura, bone, or deemed unsafe by the principal investigator
4. Patient is male or female and ≥18 years of age on the day of signing informed consent.
5. Patient must have performance status of 0-1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale and life expectancy > 3 months
6. Patient must have evaluable disease
7. Patient must have adequate organ function as indicated by the following laboratory values:

   Hematological
   * Absolute neutrophil count (ANC) ≥ 1,500 /μL
   * Platelets ≥ 100,000 /μL
   * Hemoglobin ≥ 9 g/dL

   Renal
   * Serum creatinine or calculated creatinine clearance ≤ 1.5 x upper limit of normal (ULN) OR
   * ≥ 60 mL/min for patients with creatinine levels > 1.5 x institutional ULN

   Hepatic
   * Serum total bilirubin ≤ 1.5 x ULN OR direct bilirubin ≤ ULN for patients with total bilirubin levels > 1.5 x ULN
   * Aspartate aminotransferase (AST) / serum glutamic-oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT) / serum glutamic-pyruvic transaminase (SGPT) ≤ 2.5 x ULN, ≤ 5 x ULN if liver metastasis

   Coagulation
   * Prothrombin time (PT)/International Normalized Ratio (INR) ≤ 1.2 x ULN
   * Partial thromboplastin time (PTT) ≤ 1.2 x ULN
8. Female patient of childbearing potential must have a negative serum or urine pregnancy test β-human chorionic gonadotropin (hCG) within 72 hours prior to first doses of study medication . If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
9. Female subjects of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study medication.

   Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
10. Male subjects of childbearing potential must agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
11. Patient has voluntarily agreed to participate by giving written informed consent
12. Concomitant use of bisphosphonates or nuclear factor-κB (RANK) ligand inhibitors is allowed.

EXCLUSION CRITERIA:

1. Patient who has had radiotherapy within 1 week (or unresolved radiation-related toxicities), chemotherapy within 2 weeks or 5 half-lives, whichever is longer (6 weeks for nitrosoureas, mitomycin C or bevacizumab), anti-cancer monoclonal antibody for direct anti-neoplastic treatment within 3 weeks, or who has not recovered from toxicity due to previous agents administered. If the patient has residual toxicity from prior treatment, toxicity must be ≤ Grade 1 (except for neuropathy and alopecia).
2. > 2 lines of prior chemotherapy in the metastatic setting
3. Serum lactate dehydrogenase (LDH) > 1.5x institutional ULN
4. Patients less than 2 weeks post major surgical procedure (all surgical wounds must be fully healed). For the purpose of this criterion, a major surgical procedure is defined as one requiring the administration of general anesthesia.
5. Patient is currently participating in a study with an investigational compound or device.
6. Patient has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. However, patients with CNS metastases who have completed a course of therapy would be eligible for the study provided they are clinically stable for at least 4 weeks prior to entry as defined as: (1) no evidence of new or enlarging CNS metastasis on brain imaging within 4 weeks of enrollment (2) off steroids for 2 weeks. Patients with clinically insignificant brain metastases that do not require treatment are eligible.
7. Patient has a primary central nervous system tumor
8. Patient has known hypersensitivity to the components of study drug or its analogs.
9. Patient has a history or current evidence of clinically significant heart disease including:

   * Clinically significant congestive heart failure, unstable angina pectoris,
   * Clinically significant cardiac arrhythmia,
   * Myocardial infarction during the last 6 months, and/or a current ECG tracing that is abnormal in the opinion of the treating Investigator,
   * QTc prolongation >480 msec (Bazett's Formula),
   * Congenitally long QT syndrome, and/or current anti-arrhythmic therapy
10. Patient with evidence of clinically significant bradycardia (HR <50), or a history of clinically significant bradyarrhythmias such as sick sinus syndrome, 2nd degree atrioventricular (AV) block (Mobitz Type 2), Patient with uncontrolled hypertension (≥140/90 mmHg). Patients who are controlled on antihypertensive medication will be allowed to enter the study.
11. Patient has a history or current evidence of any condition, therapy, or lab abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating investigator.
12. Patient has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
13. Patient is, at the time of signing informed consent, a regular user of any illicit drugs or had a recent history (within the last year) of drug or alcohol abuse.
14. Patient is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study
15. Patient is known to be Human Immunodeficiency Virus (HIV)-positive
16. Patient has known history of active Hepatitis A, B, or C
17. Patients who have known allergic reactions to IV contrast dye despite standard prophylaxis
18. Patients who require medications that are strong CYP3A4 inhibitors or inducers.
19. Patients who have discontinued any of these medications must have a wash-out period of at least 5 days or at least 5 half-lives of the drug (whichever is longer) prior to the first dose of dinaciclib (Refer to Appendix 2 Drugs that interact strongly with CYP3A4).
20. Patients requiring warfarin therapy are excluded, low molecular weight heparin is permitted.
21. Patient has a diagnosis of immunodeficiency or is receiving ongoing immunosuppressive therapy, including systemic or enteric corticosteroids except for non-systemically absorbed treatments (such as inhaled or topical steroid therapy for asthma, chronic obstructive pulmonary disease, allergic rhinitis). Patient must be off systemic steroid or any other form of immunosuppressive therapy within 7 days prior to first dose of trial treatment.
22. Patient is diagnosed with active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Note: replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment.
23. Patient has history of interstitial lung disease or known history of, or any evidence of active, noninfectious pneumonitis.
24. Patient has history of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or prior allogeneic bone marrow transplantation or prior solid organ transplantation.
25. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Inclusion of women and minorities:

Both men and women and members of all races and ethnic groups are eligible for this trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-12-28 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Up to 1 cycle (1 cycle is equal to 21 days)
  The MTD is determined by the number of dose-limiting toxicities reported by participants in the first cycle of treatment.
Proportion of participants with reported dose-limiting toxicities (DLTs) | Up to 1 cycle (1 cycle is equal to 21 days)
  Dose-limiting hematologic and non-hematologic toxicities classified using the CTCAE, will be based on events occurring during the first cycle of study drug administration. To be considered a dose-limiting toxicity, an adverse experience must be related to one or both of the study drugs, and must not be related to disease progression or intercurrent illnesses. Participants must receive Day 1 and Day 8 treatments of dinaciclib during the first cycle in order to be evaluable for DLTs (unless missed doses are due to toxicity).

SECONDARY OUTCOMES:
Overall Response Rate | Up to 3 years
  Overall tumor response and time to progression will be assessed using RECIST (Response Evaluation Criteria in Solid Tumors) 1.1 criteria and immune-related RECIST (irRECIST) which takes into account the clinical condition/stability of subjects in addition to tumor imaging. The rate of participants with a confirmed response classified as Complete Response (CR, iCR) (the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm) or a Partial Response (PR, iPR) (defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters or unconfirmed progressive disease (iUPD) will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: A. Jo Chien, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No